CLINICAL TRIAL: NCT05480267
Title: Unilateral Biportal Endoscopy Versus MIS-TLIF in Lumbar Spondylolisthesis: A Randomized Control Trial
Brief Title: A RCT of UBE vs. MIS-TLIF in Lumbar Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Li fangcai, Ph.D and MD., Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBE vs. MIS-TLIF
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Spondylolisthesis; Unilateral Biportal Endoscopy; Minimally Invasive Technique; Surgical Treatment
MeSH Terms: conditions — Spondylolisthesis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UBE (Experimental): The patient treated with unilateral biportal endoscopy (UBE)
  Interventions: Procedure: surgical treatment for lumbar spondylolisthesis
- MIS-TLIF (Active Comparator): The patient treated with classical minimally invasive posterior spinal interbody fusion (MIS-TLIF)
  Interventions: Procedure: surgical treatment for lumbar spondylolisthesis

INTERVENTIONS:
Procedure: surgical treatment for lumbar spondylolisthesis — There are two surgical treatments for lumbar spondylolisthesis; one is UBE, and another is MIS-TLIF

SUMMARY:
Unilateral biportal endoscopy (UBE) is a new spinal minimally invasive technique improved for the treatment of lumbar spondylolisthesis (LSP). The present study aims to establish a multicenter, large sample, randomized controlled study to explore the technical advantages and surgical indications of this new technique in the treatment of LSP by comparing with the classical minimally invasive posterior spinal interbody fusion; to compare the postoperative clinical and imaging results and analyze the surgical complications and preventive measures.

DETAILED DESCRIPTION:
Lumbar spondylolisthesis (LSP) is the most common degenerative lumbar disease in the elderly, and the severe patients need surgical treatment. The elderly are often complicated with many medical diseases and the perioperative risk is high, so minimally invasive surgery is a new direction for spinal surgeons to treat LSP. Unilateral biportal endoscopy (UBE) is a new spinal minimally invasive technique improved. The results of pilot studies showed that it had the advantages of less traumas, fewer complications, quicker recover，and the clinical and imaging outcome was remarkable. Therefore, the present study aims to establish a multicenter, large sample, randomized controlled study to explore the technical advantages and surgical indications of this new technique in the treatment of LSP by comparing with the classical minimally invasive posterior spinal interbody fusion; (2) to compare the postoperative clinical and imaging results and analyze the surgical complications and preventive measures; (3) to establish two-year follow-up to further quantify the clinical and imaging outcome of UBE. Therefore, the present study will further verify and quantify the safety and effectiveness of the UBE in the treatment of LSP on the basis of previous studies, and provide a new clinical approach for minimally invasive treatment of LSP.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spondylolisthesis,
* 40 yrs<age< 75yrs
* fusion levels <2

Exclusion Criteria:

* greater than Lenke-slivia classification III
* severe osteoporosis (t value <2.5)
* ASA 》IV

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
ODI score | 2 year postoperatively
  the D-value between the preoperative ODI score and 2-year-postoperative ODI score

CONTACTS AND LOCATIONS:
Overall Officials: Gang CHEN, MD., Principal Investigator — 2nd hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No
We have not decided when to share the plan. We plan to share it after the study completion.

REFERENCES:
- [Result] MUTCH J, WALMSLEY R. The aetiology of cleft vertebral arch in spondylolisthesis. Lancet. 1956 Jan 14;270(6907):74-7. doi: 10.1016/s0140-6736(56)92130-4. No abstract available. PMID 13287061
- [Result] Oster BA, Kikanloo SR, Levine NL, Lian J, Cho W. Systematic Review of Outcomes Following 10-Year Mark of Spine Patient Outcomes Research Trial (SPORT) for Degenerative Spondylolisthesis. Spine (Phila Pa 1976). 2020 Jun 15;45(12):820-824. doi: 10.1097/BRS.0000000000003485. PMID 32205705
- [Result] Kwon JW, Park Y, Lee BH, Yoon SR, Ha JW, Kim H, Suk KS, Moon SH, Kim HS, Lee HM. Ten-Year Outcomes of Minimally Invasive Versus Open Transforaminal Lumbar Interbody Fusion in Patients With Single-Level Lumbar Spondylolisthesis. Spine (Phila Pa 1976). 2022 Jun 1;47(11):773-780. doi: 10.1097/BRS.0000000000004334. Epub 2022 Feb 3. PMID 35125463
- [Result] Park SM, Park J, Jang HS, Heo YW, Han H, Kim HJ, Chang BS, Lee CK, Yeom JS. Biportal endoscopic versus microscopic lumbar decompressive laminectomy in patients with spinal stenosis: a randomized controlled trial. Spine J. 2020 Feb;20(2):156-165. doi: 10.1016/j.spinee.2019.09.015. Epub 2019 Sep 19. PMID 31542473
- [Result] Lightsey HM 4th, Pisano AJ, Striano BM, Crawford AM, Xiong GX, Hershman S, Schoenfeld AJ, Simpson AK. ALIF Versus TLIF for L5-S1 Isthmic Spondylolisthesis: ALIF Demonstrates Superior Segmental and Regional Radiographic Outcomes and Clinical Improvements Across More Patient-reported Outcome Measures Domains. Spine (Phila Pa 1976). 2022 Jun 1;47(11):808-816. doi: 10.1097/BRS.0000000000004333. Epub 2022 Feb 3. PMID 35125462
- [Result] Heo DH, Lee DC, Park CK. Comparative analysis of three types of minimally invasive decompressive surgery for lumbar central stenosis: biportal endoscopy, uniportal endoscopy, and microsurgery. Neurosurg Focus. 2019 May 1;46(5):E9. doi: 10.3171/2019.2.FOCUS197. PMID 31042664
- See also: Comparative analysis of three types of minimally invasive decompressive surgery for lumbar central stenosis — http://www.ncbi.nlm.nih.gov/pubmed/31042664
- See also: ALIF Demonstrates Superior Segmental and Regional Radiographic Outcomes and Clinical Improvements Across More Patient-reported Outcome Measures — http://www.ncbi.nlm.nih.gov/pubmed/35125462
- See also: Biportal endoscopic versus microscopic lumbar decompressive laminectomy in patients with spinal stenosis: a randomized controlled trial — http://www.ncbi.nlm.nih.gov/pubmed/31542473